CLINICAL TRIAL: NCT07215442
Title: Skin Temperature Perception and Prosthetic Thermoregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn K. Klute, PhD, Director, CLiMB, VA Puget Sound Health Care System
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1587700
Record Dates: First submitted 2025-09-26; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Lower Limb Amputation Below Knee; Diabetes (DM); Skin Temperature Change; Vascular Reactivity
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individuals without a diagnosis of diabetes (Other)
  Interventions: Other: Warming stimulus starting at 30 C initial temperature; Other: Warming stimulus starting at 32 C initial temperature; Other: Warming stimulus starting at 34 C initial temperature; Other: Warming stimulus starting at 35 C initial temperature; Other: Cooling stimulus starting at 30 C initial temperature; Other: Cooling stimulus starting at 32 C initial temperature; Other: Cooling stimulus starting at 34 C initial temperature; Other: Cooling stimulus starting at 35 C initial temperature
- Individuals with diabetes (Other)
  Interventions: Other: Warming stimulus starting at 30 C initial temperature; Other: Warming stimulus starting at 32 C initial temperature; Other: Warming stimulus starting at 34 C initial temperature; Other: Warming stimulus starting at 35 C initial temperature; Other: Cooling stimulus starting at 30 C initial temperature; Other: Cooling stimulus starting at 32 C initial temperature; Other: Cooling stimulus starting at 34 C initial temperature; Other: Cooling stimulus starting at 35 C initial temperature
- Individuals with lower limb amputations of diabetic etiology (Other)
  Interventions: Other: Warming stimulus starting at 30 C initial temperature; Other: Warming stimulus starting at 32 C initial temperature; Other: Warming stimulus starting at 34 C initial temperature; Other: Warming stimulus starting at 35 C initial temperature; Other: Cooling stimulus starting at 30 C initial temperature; Other: Cooling stimulus starting at 32 C initial temperature; Other: Cooling stimulus starting at 34 C initial temperature; Other: Cooling stimulus starting at 35 C initial temperature
- Individuals with lower limb amputations of non-diabetic etiologies (Other)
  Interventions: Other: Warming stimulus starting at 30 C initial temperature; Other: Warming stimulus starting at 32 C initial temperature; Other: Warming stimulus starting at 34 C initial temperature; Other: Warming stimulus starting at 35 C initial temperature; Other: Cooling stimulus starting at 30 C initial temperature; Other: Cooling stimulus starting at 32 C initial temperature; Other: Cooling stimulus starting at 34 C initial temperature; Other: Cooling stimulus starting at 35 C initial temperature

INTERVENTIONS:
Other: Warming stimulus starting at 30 C initial temperature — A warming stimulus starting at 30 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 42 C was reached.
Other: Warming stimulus starting at 32 C initial temperature — A warming stimulus starting at 32 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 42 C was reached.
Other: Warming stimulus starting at 34 C initial temperature — A warming stimulus starting at 34 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 42 C was reached.
Other: Warming stimulus starting at 35 C initial temperature — A warming stimulus starting at 35 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 42 C was reached.
Other: Cooling stimulus starting at 30 C initial temperature — A cooling stimulus starting at 30 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 18 C was reached.
Other: Cooling stimulus starting at 32 C initial temperature — A cooling stimulus starting at 32 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 18 C was reached.
Other: Cooling stimulus starting at 34 C initial temperature — A cooling stimulus starting at 34 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 18 C was reached.
Other: Cooling stimulus starting at 35 C initial temperature — A cooling stimulus starting at 35 C initial temperature was applied at a rate of 0.2 C/second until the participant perceived the stimulus or the termination temperature of 18 C was reached.

SUMMARY:
To protect against excessive body temperatures, local thermoregulatory mechanisms include temperature sensory nerves (responsive to warm or cool stimuli) and vasomotors (muscles that constrict or dilate blood vessels). When the temperature changes occur, the temperature sensory nerves will detect "warm" or "cool" and communicate this sensation to the brain. This is called perceiving a sensation and will often elicit a behavioral change, such as donning additional clothes or moving to a different environment. Simultaneously, vasomotors will dilate or constrict to promote or prevent heat dissipation to the environment, respectively. As skin temperatures increase, perspiration may provide some thermal relief through evaporative cooling. However, the prostheses worn by individuals with lower limb amputations are impermeable to moisture and prevent evaporative cooling. Prosthetic materials are also excellent thermal insulators, contributing to skin temperature increases. Thermoregulation problems are compounded by diabetes, a common co-morbidity of many who experience lower limb amputation. For those who wear lower limb prostheses, many endure thermal discomfort.

This research explores the relationship between skin temperature, perception, and thermoregulation. The investigators aim to discover the temperature at which individuals with lower limb amputation perceive warm and cool stimuli. The investigators also aim to discover the vascular response that occurs when temperature changes are perceived. The goals are to determine temperature sensation thresholds of the lower limb, vascular reactivity, and the effect of diabetes and amputation.

DETAILED DESCRIPTION:
This study will include four groups of participants including individuals with diabetes, individuals without a diagnosis of diabetes, individuals with lower limb amputations of diabetic etiology, and individuals with lower limb amputations of non-diabetic etiologies.

To measure temperature perception, a thermode (a temperature changing device about the size of a coffee cup) will be placed on the lower leg of each participant. The thermode also included a laser Doppler flow meter, embedded in the center of the thermode, to measure blood flow in response to changes in skin temperature. The experimental protocol begins with the thermode set for 3 minutes at 30 °C, 32 °C, 34 °C, and 35 °C (random order). The temperature will then be either increased or decreased at a slow rate of 0.2 °C/sec until the participant perceives either a warming or cooling sensation. The analysis plan includes determining the threshold at which a temperature change was perceived relative to each initial temperature, whether there are differences in blood flow (vascular reactivity) when thermal stimuli are detected, and these measurements are altered by diabetes or amputation.

The general hypotheses are that these populations will have (1) different warm and cool temperature perception thresholds depending on the initial skin temperature and (2) different changes in skin blood flow as a function of their temperature perception thresholds.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Able to ambulate without upper extremity aids
* Able to attend study visits
* Able to sense a Semmes-Weinstein 5.07 monofilament applied to proximal lateral aspect of test limb calf
* Cognitively aware Additional Inclusion Criteria for Individuals with Lower Limb Amputation
* Have been fit with a prosthesis
* Have used a prosthesis for at least six months
* Wear the prosthesis for at least four hours per day by self-report

Exclusion Criteria for Individuals with Lower Limb Amputation:

- Have no residual limb ulcers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

PRIMARY OUTCOMES:
Thermal perception threshold | Day 1
  The thermal perception threshold is the difference between the initial temperature and the temperature at which the participant detected the thermal stimulus
Skin blood flow difference | Day 1
  The skin blood flow difference is the difference between the skin blood flow at the initial temperature and the skin blood flow at the temperature at which the participant detected a thermal stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, Washington, United States